CLINICAL TRIAL: NCT04333212
Title: Human Papillomavirus Detection and Genotyping by DR. HPV Genotyping IVD Kit in Exfoliated Cells of the Uterine Cervix
Brief Title: HPV Genotyping by DR. HPV Genotyping in Vitro Diagnostic Device (IVD) Kit in Exfoliated Cells of the Uterine Cervix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Dr. Chip Biotechnology Incorporation (Other)
Responsible Party: Principal Investigator, TING-CHANG CHANG, Professor and Chairperson, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MA1103L9
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Cervical Intraepithelial Neoplasia; Human Papillomavirus Infection; HPV Infection
MeSH Terms: conditions — Uterine Cervical Dysplasia; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study arm (Other): We projected a total of 1,100 study cases, which encompassed 100 cases of women with no intraepithelial lesion or malignancy (NILM) cytology, 300 cases of ASCUS, 300 cases of low grade squamous intraepithelial lesion (LSIL) and 400 cases high grade squamous intraepithelial lesion (HSIL) in cervical cytology.
  Interventions: Device: DR. Chip HPV genotyping IVD kit

INTERVENTIONS:
Device: DR. Chip HPV genotyping IVD kit — HPV typing by gene chip

SUMMARY:
High-risk type human papillomavirus (HPV) is the known etiological agent of cervical cancer. HPV testing and risk stratification by genotyping has been recognized as an effective cervical screening program. A chip for HPV DNA typing based on type-specific polymerase chain reaction (PCR), DR. HPV Genotyping IVD Kit (HPV-27) was developed for genotyping of 27 common HPV types including all high-risk types. We studied its agreement, sensitivity, and specificity compared to DNA sequencing as the gold standard.

DETAILED DESCRIPTION:
High-risk type human papillomavirus (HPV) is the known etiological agent of cervical cancer. HPV testing and risk stratification by genotyping has been recognized as an effective cervical screening program. HPV detection is also applied for triage of atypical squamous cells of undetermined significance and follow-up after treatment for cervical neoplasms. A chip for HPV DNA typing based on type-specific polymerase chain reaction (PCR), DR. HPV Genotyping IVD Kit (HPV-27) was developed for genotyping of 27 common HPV types including all high-risk types. We studied its agreement, sensitivity, and specificity compared to DNA sequencing as the gold standard.

One-thousand one-hundred and three (1103) subjects were enrolled between December 2012 and December 2013 from Linkou Chang Gung Memorial Hospital, Mackay Memorial Hospital, Changhua Christian Hospital, and Cathay General Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. 21-65 y/o female with sexual exposure
2. Written informed consent
3. Either one of the following conditions:

3a. No previous history of abnormal cervical cytology or abnormal histology for women enrolled in no intraepithelial lesion or malignancy (NILM) group 3b. Abnormal cervical cytology other than atrophic change, reactive change or glandular cells favored of the endometrial origin

Exclusion Criteria:

1. Current pregnancy
2. Previous total hysterectomy
3. Cervicovaginal infection required treatment
4. Received cervical ablative therapy within 1 year

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — HPV detection and typing for exfoliated cervical cells
Enrollment: 1103 (Actual)
Dates: Start 2012-12-12 (Actual); Primary Completion 2013-12-30 (Actual); Study Completion 2014-07-08 (Actual)

PRIMARY OUTCOMES:
Agreement | within one week after sample collected by a study physician
  agreement, sensitivity, and specificity compared to DNA sequencing

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - Changhua Christian Hospital, Changhua
  - Mackay Memorial Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
For clinical trial participation
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 months after accepting for report publication
Access Criteria: to the public